CLINICAL TRIAL: NCT04922125
Title: Impact of Pulse Processing on Feelings of Appetite and Satiety
Brief Title: Food Structure of Pulses and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Katharina Pälchen, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UCopenhagen 514-0254/21-5000
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: A single-blind, randomised crossover design with one arm.
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse flour (Experimental): Puree produced from pulse flours and with added oil and herbs/spices. To standardize test products on textural aspects, different levels of thickener will be added. All test products will be produced in the Future Consumer Lab at the Department of Food Science at the University of Copenhagen prior to the appetite test days. Pulse flour will be produced in the food-grade laboratory environment at the Department of Food Design and Consumer behavior and dried prior to use.
  Interventions: Combination Product: Pulse flour
- Pre-processed pulse flour (Experimental): Puree produced from pre-processed pulse flour with different structural aspects and with added oil and herbs/spices. To standardize test products on textural aspects, different levels of thickener will be added. All test products will be produced in the Future Consumer Lab at the Department of Food Science at the University of Copenhagen prior to the appetite test days. Pulse flour will be produced in the food-grade laboratory environment at the Department of Food Design and Consumer behavior and dried prior to use.
  Interventions: Combination Product: Pre-processed pulse flour

INTERVENTIONS:
Combination Product: Pulse flour — Traditionally processed pulse flour in vitro digestion conditions were related to potentially influence appetite sensations.
  Arms: Pulse flour
Combination Product: Pre-processed pulse flour — Pre-processing of pulse flour was related to altered in vitro digestion conditions and thus suggested to potentially influence appetite sensations.
  Arms: Pre-processed pulse flour

SUMMARY:
Diets containing (whole) pulses have been associated with the potential to increase satiety (and acute food intake). In vitro digestion studies of pulses have shown that (thermal) processing has the potential to modulate macronutrient digestion kinetics. Changes in food (micro)strucutral properties have been identified to retard nutrient release, with a possible effect on appetite sensations. Based on distinct in vitro digestion behaviour, two differently processed pulse meals were chosen to be investigated in humans with the aim to confirm in vitro findings and gain a mechanistic understanding of the influence of structural aspects of pulses on appetite sensations.

ELIGIBILITY:
Inclusion Criteria:

* BMI (between 18 and 30 kg/m2)
* Healthy men
* Age between 18-45
* Regular breakfast eaters (≥ 4 times a week)
* No allergies

Exclusion Criteria:

* Chronic diseases (diabetes, cardiovascular diseases, or other metabolic diseases that could affect the study)
* Use of daily prescription medicine
* Use of dietary supplements that could affect appetite (used within the last month up to or during the study)
* Smoking or use of any nicotine product (used daily within the last three months up to or during the study)
* Over 10 h of strenuous physical activity per week
* Participation in other clinical studies (participation within the last month up to the study or during the study)
* Food allergies
* Weight change of more than ±3 kg from screening until the trial will be completed
* Inability to comply with the procedures required by the study (including an 8-10 h fast before the trial days).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Self-reported appetite assessment throughout the appetite test days | 2.5 hours
  Visual analogue scales (VAS) will be measuring differences in perception of satiety, fullness, hunger and predicted prospective food consumption between the experimental condition compared to the control condition, with VAS 0-100 mm with 0 indicating no hunger or perceived ability to consume food / no satiety or no fullness)

SECONDARY OUTCOMES:
Secondary Energy Intake (kJ) of ad libitum meal | 30 min
  Differences in (secondary) energy intake after the test-meals at the ad libitum meal will be compared to the control condition
Satiety quotient (SQ) | 30 min
  Visual analogue scales (VAS) will be measuring differences in SQ consumption before and after the experimental condition compared to the control condition (0-100 mm with 0 indicating no hunger or perccieved ability to consume food / no satiety or no fullness)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science/ Section for Food Design and Consumer Behaviour, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No